CLINICAL TRIAL: NCT06471166
Title: The Effect of Different Treatment Modalities of Tubal Ectopic Pregnancy on Ovarian Reserve: a Prospective Cohort Study
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Andro Bahgat Heshmat, Resident, Assiut University
Other Study IDs: Ectopic pregnancy
Record Dates: First submitted 2024-06-18; First posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Ectopic Pregnancy
MeSH Terms: conditions — Pregnancy, Ectopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (6):
- Conservative management
  Interventions: Diagnostic Test: Amh hormone
- Medical treatment
  Interventions: Diagnostic Test: Amh hormone
- Surgical treatment (Open or laparoscopic salpingectomy)
  Interventions: Diagnostic Test: Amh hormone
- Surgical treatment after failed medical treatment (Open or laparoscopic salpingectomy)
  Interventions: Diagnostic Test: Amh hormone
- Conservative surgical treatment (salpingotomy, salpingostomy, tubal milking)
  Interventions: Diagnostic Test: Amh hormone
- Conservative surgical treatment after failed medical treatment
  Interventions: Diagnostic Test: Amh hormone

INTERVENTIONS:
Diagnostic Test: Amh hormone — Ovarian reserve

SUMMARY:
Detect the effect of different treatment modalities of tubal ectopic pregnancy on ovarian reserve

ELIGIBILITY:
Inclusion Criteria:

* The study will include patients aged 18-44 years with known diagnosis or suspicion of diagnosis of tubal ectopic pregnancy (abnormal doubling rates of their b-HCG levels as well as ultrasonographically identified or unidentified gestational sacs outside the uterus)
* Included patients must have capacity to provide informed consent. Given the potential emergent nature of presentation, women will not be recruited if fully informed consent could be compromised due to a highly distressed emotional state or significant hemorrhage necessitating the need for urgent surgery

Exclusion Criteria:

1. The use of hormonal contraceptives within two months of enrolment
2. If other surgery was conducted at the time of salpingectomy.
3. If a woman was pregnant at follow up visit for AMH measurement
4. History of previous surgeries of fallopian tubes and/or ovaries

Ages: 18 Years to 44 Years | Sex: Female
Age Groups: Adult
Study Population: Women's Health Hospital, Department of Obstetrics and Gynecology, Faculty of Medicine, Assiut University
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-07-10 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-10 (Estimated)

PRIMARY OUTCOMES:
Change in levels of AMH pre and post treatment | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt